CLINICAL TRIAL: NCT03596242
Title: Short Message Service System for Patients With Uncontrolled Hypertension
Brief Title: SMS System for Patients With Uncontrolled Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00051763; 5UL1TR001420-03 (NIH)
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-03

CONDITIONS: Hypertension
Keywords: high blood pressure; SMS; text messaging; monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Blood Pressure Monitoring by Short Message Service (SMS) (Experimental): Will receive the text message intervention and will be provided with a blood pressure cuff in addition to standard blood pressure control education received at clinic visits
  Interventions: Other: SMS System; Behavioral: blood pressure control education
- Usual Care Plus Standard Blood Pressure Monitoring (Active Comparator): Will receive standard blood pressure care and education, as well as a blood pressure cuff at their clinic visits
  Interventions: Behavioral: blood pressure control education

INTERVENTIONS:
Other: SMS System — Participants will receive usual care +SMS texting and phone calls to monitor their blood pressure and medication adherence
  Arms: High Blood Pressure Monitoring by Short Message Service (SMS)
Behavioral: blood pressure control education — standard blood pressure control education given during visits

SUMMARY:
This is a pilot study to determine the potential of utilizing Short Message Service (SMS) messaging to improve health outcomes for patients with uncontrolled hypertension receiving care from the Outpatient Internal Medicine Clinic at Wake Forest Baptist Hospital.

DETAILED DESCRIPTION:
The pilot will evaluate the feasibility of implementing a Short Message Service (SMS) system and Home Blood Pressure Measurements (HBPM) in the Outpatient Internal Medicine (OPD) clinic at Wake Forest Baptist Hospital. Implementing a new short text messaging service will improve the health delivery system in three ways. 1) Increasing patient engagement: SMS and HBPM require an active commitment by the patients themselves in their medical care and results in a marked improvement in the adherence to medication. High adherence to home blood pressure (BP) measurements has also been reported to improve BP control. 2) Supporting patients outside of the office visits by identifying and resolving barriers to medication adherence earlier on (i.e. if patients are unable to get their prescriptions or are having significant side effects). 3) Adopting clinical guidelines to improve BP control in a vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with hypertension
* 18 and older
* stage 2 hypertension or greater systolic blood pressure [(SBP)>140 and diastolic blood pressure (DBP) >90] who are receiving antihypertensive treatment.

Exclusion Criteria:

* Pregnancy
* end-stage renal disease (on hemodialysis or peritoneal dialysis)
* hospice or nursing home care
* dementia
* Patients who do not have a phone with Short Message Service (SMS) capabilities will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Campos, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lauffenburger JC, Choudhry NK. Text Messaging and Patient Engagement in an Increasingly Mobile World. Circulation. 2016 Feb 9;133(6):555-6. doi: 10.1161/CIRCULATIONAHA.116.021182. Epub 2016 Jan 14. No abstract available. PMID 26769741
- [Derived] Campos CL, Jones D, Snively BM, Rocco M, Pedley C, Atwater S, Moore JB. Text Messaging and Home Blood Pressure Monitoring for Patients with Uncontrolled Hypertension: Proposal for a Feasibility Pilot Randomized Controlled Trial. JMIR Res Protoc. 2021 May 14;10(5):e18984. doi: 10.2196/18984. PMID 33988513

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Blood Pressure Monitoring by Short Message Service (SMS) | Usual Care Plus Standard Blood Pressure Monitoring
Started | 12 | 12
Completed | 10 | 10
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- High Blood Pressure Monitoring by SMS: Will receive the text message intervention and will be provided with a blood pressure cuff in addition to standard blood pressure control education received at clinic visits
  SMS System: Participants will receive usual care +SMS texting and phone calls to monitor their blood pressure and medication adherence
  blood pressure control education: standard blood pressure control education given during visits
- Total: Total of all reporting groups
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (13.0) | 53.6 (11.1) | 55.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Screened
Time Frame: during screening period, about 6 months
Measure: Number; unit: participants
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 12 | 12
participants | 12 | 12

2. Primary Outcome: Number of Subjects Enrolled
Time Frame: during baseline period, about 4 months
Measure: Number; unit: participants
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 12 | 12
participants | 12 | 12

3. Primary Outcome: Number of Subjects Who Refuse Participation
Description: number of participants who refuse to participate at the time of recruitment and the reason why
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

4. Primary Outcome: Number of Subjects Excluded Without SMS Capability
Description: Number of vulnerable subjects screened but excluded because they did not own a phone with SMS capability.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

5. Primary Outcome: Proportion of Participants Continuing myHealth
Description: the proportion of participants who continue to use the myHealth tool per month through three months will be tracked for the intervention
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

6. Primary Outcome: Number of Participants Who Responded to SMS With At Least One Home BP Measurement
Time Frame: up to 12 weeks
Population: This was only measured in the "High Blood Pressure Monitoring by SMS" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | High Blood Pressure Monitoring by SMS
Number analyzed (Participants) | 12
Participants | 8

7. Primary Outcome: SMS Participation
Description: The number of patients who participate in SMS will be recorded
Time Frame: up to 12 weeks
Population: This outcome was only measured in the "High Blood Pressure Monitoring by SMS" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | High Blood Pressure Monitoring by SMS
Number analyzed (Participants) | 12
Participants | 12

8. Primary Outcome: System Usability Scale (SUS)
Description: Participants will complete the SUS in person on an I-Pad or over the phone. The SUS yields a single score on a scale of 0-100. A SUS score above a 68 would be considered above average (better) usability.
Time Frame: Week 12
Population: Only 8 people in the SMS arm completed the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Blood Pressure Monitoring by SMS
Number analyzed (Participants) | 8
score on a scale | 92.25 (121.7)

9. Secondary Outcome: Medication Adherence
Description: The number of patients who demonstrate medication compliance via SMS will be recorded.
Time Frame: up to 12 weeks
Population: Information not obtained for this outcome measure
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Medication Adherence Questionnaire
Description: Score ranges from 0 to 10 with higher score denoting better medication adherence.
Time Frame: baseline, week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 10 | 10
score on a scale
  baseline | 2.17 (0.93) | 2.02 (0.7)
  Week 12 | 0.93 (1.2) | 1.8 (2.09)

11. Secondary Outcome: Monitoring of SBP
Description: Changes in values of Systolic blood pressure (SBP) received via SMS will be recorded
Time Frame: baseline and 12 weeks
Population: Only 8/12 responded with their SBP in the "High Blood Pressure Monitoring by SMS" and 10/12 responded with their SBP in the "Usual Care Plus Standard Blood Pressure Monitoring".
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 8 | 10
mmHg | 15 (2.8) | 13 (3.4)

12. Secondary Outcome: Monitoring of DBP
Description: Changes in values of Diastolic blood pressure (DBP) received via SMS will be recorded
Time Frame: baseline and 12 weeks
Population: Only 8/12 responded with their DBP in the "High Blood Pressure Monitoring by SMS" and only 10/12 responded with their DBP in the "Usual Care Plus Standard Blood Pressure Monitoring"
Measure: Mean (Standard Deviation); unit: change in mmHg
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 8 | 10
change in mmHg | 10 (3.2) | 8 (2.0)

13. Secondary Outcome: Initial and Follow up BP in Office
Description: Number of participants to attended both initial and follow up blood pressure (systolic and diastolic) visits will be recorded.
Time Frame: baseline/day 0 and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 10 | 10
Participants
  Baseline | 10 | 10
  Week 12 | 10 | 10

14. Secondary Outcome: Number of Participants Considered No-Shows at Clinic Visits
Description: No-show rate at 3 months' follow-up (f/u) clinic visits. If participants fail to come to their f/u visits within 7 days of their scheduled follow-up appointment, they will be considered as "no- shows".
Time Frame: week 12
Measure: Number; unit: participants
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 11 | 11
participants | 1 | 1

15. Secondary Outcome: Coordinator Time
Description: The time spent by the coordinator on study related patient activities will be recorded
Time Frame: up to 12 weeks
Population: Measure data not collected
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: baseline through week 12
Arm/Group | High Blood Pressure Monitoring by SMS | Usual Care Plus Standard Blood Pressure Monitoring
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT03596242/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT03596242/ICF_000.pdf